CLINICAL TRIAL: NCT01531153
Title: Cognitive Enhancement as a Target for Cocaine Pharmacotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1007007119; R01DA029577 (NIH)
Record Dates: First submitted 2011-12-07; First posted 2012-02-10 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Addiction
Keywords: Cocaine use decreases, increases or stays the same
MeSH Terms: conditions — Behavior, Addictive | interventions — Galantamine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar Pill (Active Comparator): Sugar Pill will be compared with the active medication Galantamine
  Interventions: Drug: Placebo
- Galantamine (Active Comparator): Comparing the active medication with the placebo medication to see if the self administration cocaine decreases.
  Interventions: Drug: Galantamine

INTERVENTIONS:
Drug: Galantamine — 8mg or 16mg
  Other Names: Razadyne; Razadyne ER
  Arms: Galantamine
Drug: Placebo — Placebo dose.
  Other Names: Sugar Pill
  Arms: Sugar Pill

SUMMARY:
Specific Aim #1: To determine if galantamine (8 or 16 mg/day) is more effective than placebo in reducing cocaine use as measured by cocaine urine results and self-report days of use.

Specific Aim # 2: To determine if galantamine (8 or 16 mg/day) is more effective than placebo in improving attention, assessed with the Rapid Visual Information Processing (RVIP) and the Simple Reaction Time (SRT) tests Specific Aim # 3: To determine if improvement in attention during the first four weeks of treatment will mediate galantamine's efficacy in reducing cocaine use.

DETAILED DESCRIPTION:
This will be a double-blind, placebo-controlled, randomized clinical trial. One hundred and twenty cocaine-dependent men and women will be randomized to one of three treatment groups: placebo (n=40), 8 mg/day (n=40), and 16 mg/day (n=40) of extended release (ER) galantamine. An urn randomization will be used to balance the groups for gender, severity of cocaine use (measured by days of cocaine use), baseline cognitive functioning [determined via the Shipley Institute of Living Scale (SILS)], and smoking status. Gender and severity of cocaine use have been shown to predict treatment responses in cocaine users (76). Similarly, balancing the treatment groups for baseline cognitive functioning, assessed with the SILS scores, will minimize the influence of baseline differences on cognitive outcomes (77, 78). Smoking status is also an important baseline variable, given galantamine's actions on nicotinic receptors and its potential efficacy for smoking cessation (65). The initial dose of galantamine will be 8 mg/day as a single dose, as recommended for clinical use. For those assigned to 16 mg/day, the dose of galantamine will be increased to 16 mg at the end of week 4. Treatment groups will remain on their full dosage through week 13. All participants will receive contingency management (CM) targeting treatment compliance. In three previous cocaine pharmacotherapy trials using bupropion, desipramine or levodopa, medication efficacy on cocaine use was evident only when medications were combined with CM, but not with standard care (79-81). These findings provide a strong rationale for using CM in our clinical trial.

Recruitment is continuing. This protocol was amended as of May 2014 to come to one dispensing visit and up too, two clinic visits. The payment has changed from gift cards to cash. This change should help increase the number of completers.

Currently there are 40 completers with 9 active and 6 in follow up phase. The follow up phase ended June 2016. Currently in analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females, between the ages of 18 and 60
2. Are using cocaine more than once per week in the previous 30 days, provide a cocaine-positive urine specimen at screening, and fulfill criteria for current cocaine dependence according to DSM-IV
3. For women of child-bearing age, have a negative pregnancy test at screening, agree to adequate contraception to prevent pregnancy, and agree to have monthly pregnancy tests
4. Are fluent in English and have a 6th grade or higher reading level; AND
5. Can commit to at least 13 weeks of treatment and are willing to be randomized to treatment

Exclusion Criteria:

1. Meet DSM-IV psychiatric classifications for lifetime schizophrenia or bipolar disorder, or have a depressive or anxiety disorder with current use of a prescribed psychotropic medication that cannot be discontinued
2. Current DSM-IV diagnosis of drug or alcohol dependence (other than cocaine, or tobacco)
3. Demonstrate significant medical conditions, including asthma or chronic obstructive lung disease, history or current gastrointestinal ulcer, hepatic or renal deficit and cardiac rhythm disturbances or any other medical conditions that the study physician deems contraindicated for galantamine treatment
4. Use of other medications including:

   * drugs that slow heart rate (e.g., beta-blockers), which may increase the risk of bradycardia and atrioventricular (AV) block and
   * non-steroidal anti-inflammatory drugs (NSAIDs); increased potential for developing ulcers/active or occult gastrointestinal bleeding
5. Have a screening liver function test (AST or ALT) greater than 3 times normal; OR
6. Known allergy or adverse reaction to galantamine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2011-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D., Ph.D., Principal Investigator — Yale University
Locations (1):
- Department of Veterans Affairs, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Sugar Pill will be compared with the active medication Galantamine
  Placebo: Placebo dose.
- Galantamine 8mg: Comparing the active medication with the placebo medication to see if the self administration cocaine decreases.
  Galantamine: 8mg
- Galantamine 16mg: Comparing the active medication with the placebo medication to see if the self administration cocaine decreases.
  Galantamine: 16mg
Period: Overall Study
Arm/Group | Placebo | Galantamine 8mg | Galantamine 16mg
Started | 32 | 31 | 30
Completed | 22 | 22 | 15
Not Completed | 10 | 9 | 15
Not completed — Withdrawal by Subject | 10 | 9 | 15

BASELINE CHARACTERISTICS:
Population: A total of 95 people consented, but only 93 were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Galantamine 8mg | Galantamine 16mg | Total
Number analyzed (Participants) | 32 | 31 | 30 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (7.2) | 47.4 (6.8) | 43.3 (8.3) | 46.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 9 | 30
  Male | 20 | 22 | 21 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 25 | 21 | 16 | 62
  Caucasian | 3 | 4 | 5 | 12
  Hispanic | 3 | 3 | 9 | 15
  Multiracial | 1 | 3 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 31 | 30 | 93
Marital Status [Count of Participants; unit: Participants]
  Married | 29 | 26 | 24 | 79
  Not Married | 3 | 5 | 6 | 14
Employment [Count of Participants; unit: Participants]
  Working | 7 | 6 | 8 | 21
  Not Working | 24 | 25 | 20 | 69
Education [Count of Participants; unit: Participants]
  Some College or More | 9 | 3 | 8 | 20
  High School | 15 | 17 | 16 | 48
  Less than High School | 8 | 11 | 6 | 25
Baseline Urine Positive [Count of Participants; unit: Participants]
  Cocaine | 29 | 23 | 27 | 79
  Benzodiazepines | 1 | 1 | 0 | 2
  Marijuana | 4 | 10 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Urine Toxicology
Description: Presented are the average number of urine samples positive for cocaine over 12 weeks. This outcome was corrected from the protocol registration when the study data were entered.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: average cocaine positive urine samples
Arm/Group | Placebo | Galantamine 8mg | Galantamine 16mg
Number analyzed (Participants) | 26 | 24 | 22
average cocaine positive urine samples | 16.1 (8.0) | 17 (9.4) | 14.9 (8.5)

2. Secondary Outcome: Heart Rate
Description: Pulse
Time Frame: once a day for up to two days over 12 Weeks
Population: Summary data for only those measured at each week are presented (per protocol).
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 26 | 24 | 26
beats per minute (bpm)
  Week 1 | 78.85 (12.67) | 77.76 (9.24) | 75.01 (9.31)
  Week 2: number analyzed (Participants) | 25 | 21 | 26
  Week 2 | 80.24 (13.61) | 79.74 (10.62) | 77.13 (10.62)
  Week 3: number analyzed (Participants) | 24 | 20 | 26
  Week 3 | 78.68 (11.03) | 80.42 (8.15) | 74.98 (10.86)
  Week 4: number analyzed (Participants) | 24 | 18 | 24
  Week 4 | 82.35 (11.18) | 77.83 (7.56) | 74.84 (8.52)
  Week 5: number analyzed (Participants) | 23 | 17 | 24
  Week 5 | 80.91 (10.59) | 78.82 (9.25) | 76.72 (9.68)
  Week 6: number analyzed (Participants) | 23 | 17 | 23
  Week 6 | 80.44 (11.17) | 75.55 (10.08) | 75.80 (10.08)
  Week 7: number analyzed (Participants) | 22 | 16 | 23
  Week 7 | 78.65 (13.04) | 80.50 (9.03) | 76.48 (10.76)
  Week 8: number analyzed (Participants) | 21 | 16 | 22
  Week 8 | 82.73 (12.34) | 77.46 (10.46) | 78.56 (10.02)
  Week 9: number analyzed (Participants) | 22 | 16 | 22
  Week 9 | 80.59 (11.91) | 81.31 (9.81) | 78.09 (10.15)
  Week 10: number analyzed (Participants) | 22 | 16 | 22
  Week 10 | 80.03 (13.02) | 81.28 (10.11) | 80.02 (12.00)
  Week 11: number analyzed (Participants) | 22 | 15 | 22
  Week 11 | 82.90 (10.98) | 80.51 (11.16) | 80.02 (12.15)
  Week 12: number analyzed (Participants) | 21 | 15 | 22
  Week 12 | 81.07 (10.49) | 76.33 (7.47) | 77.38 (12.60)

3. Secondary Outcome: Blood Pressure- Systolic
Description: Blood Pressure is taken for safety reasons
Time Frame: 2 times a week for 12 weeks
Population: Data are reported for those that were measured at each assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 26 | 24 | 26
mmHg
  Week 1 Time 1: number analyzed (Participants) | 26 | 24 | 24
  Week 1 Time 1 | 133.62 (14.01) | 127.75 (11.69) | 132.21 (13.68)
  Week 1 Time 2: number analyzed (Participants) | 24 | 20 | 25
  Week 1 Time 2 | 132.04 (14.27) | 125.70 (16.11) | 136.68 (16.46)
  Week 2 Time 1: number analyzed (Participants) | 25 | 21 | 26
  Week 2 Time 1 | 132.92 (14.89) | 125.62 (12.58) | 130.69 (13.56)
  Week 2 Time 2: number analyzed (Participants) | 24 | 20 | 24
  Week 2 Time 2 | 128.46 (12.46) | 129.65 (14.76) | 130.21 (16.53)
  Week 3 Time 1: number analyzed (Participants) | 24 | 19 | 26
  Week 3 Time 1 | 132.29 (13.81) | 123.05 (13.19) | 130.58 (17.35)
  Week 3 Time 2: number analyzed (Participants) | 22 | 16 | 23
  Week 3 Time 2 | 129.14 (16.10) | 131.50 (15.47) | 129.00 (28.65)
  Week 4 Time 1: number analyzed (Participants) | 24 | 17 | 24
  Week 4 Time 1 | 129.42 (15.34) | 131.47 (13.86) | 131.46 (12.55)
  Week 4 Time 2: number analyzed (Participants) | 23 | 15 | 23
  Week 4 Time 2 | 130.22 (15.13) | 130.40 (12.87) | 131.00 (13.16)
  Week 5 Time 1: number analyzed (Participants) | 23 | 17 | 24
  Week 5 Time 1 | 132.30 (17.50) | 133.12 (14.80) | 136.58 (14.83)
  Week 5 Time 2: number analyzed (Participants) | 21 | 17 | 22
  Week 5 Time 2 | 134.67 (16.21) | 128.47 (19.13) | 133.27 (15.71)
  Week 6 Time 1: number analyzed (Participants) | 23 | 16 | 23
  Week 6 Time 1 | 131.04 (17.66) | 125.94 (15.28) | 132.26 (17.56)
  Week 6 Time 2: number analyzed (Participants) | 22 | 14 | 23
  Week 6 Time 2 | 135.23 (16.01) | 124.21 (10.53) | 132.96 (10.45)
  Week 7 Time 1: number analyzed (Participants) | 22 | 16 | 23
  Week 7 Time 1 | 133.68 (12.44) | 121.50 (15.84) | 128.96 (15.62)
  Week 7 Time 2: number analyzed (Participants) | 22 | 15 | 22
  Week 7 Time 2 | 133.82 (14.32) | 125.27 (15.40) | 129.86 (12.87)
  Week 8 Time 1: number analyzed (Participants) | 21 | 16 | 22
  Week 8 Time 1 | 136.43 (19.92) | 129.56 (15.18) | 134.09 (17.12)
  Week 8 Time 2: number analyzed (Participants) | 20 | 14 | 21
  Week 8 Time 2 | 132.95 (17.00) | 133.00 (15.96) | 134.76 (14.74)
  Week 9 Time 1: number analyzed (Participants) | 22 | 15 | 22
  Week 9 Time 1 | 140.95 (43.91) | 121.93 (13.05) | 135.32 (14.36)
  Week 9 Time 2: number analyzed (Participants) | 21 | 14 | 22
  Week 9 Time 2 | 130.29 (19.31) | 130.43 (14.48) | 133.50 (17.32)
  Week 10 Time 1: number analyzed (Participants) | 22 | 16 | 21
  Week 10 Time 1 | 136.95 (16.85) | 127.00 (14.41) | 131.05 (15.08)
  Week 10 Time 2: number analyzed (Participants) | 21 | 14 | 21
  Week 10 Time 2 | 132.52 (13.13) | 121.07 (19.86) | 128.00 (15.70)
  Week 11 Time 1: number analyzed (Participants) | 22 | 14 | 21
  Week 11 Time 1 | 133.86 (14.23) | 125.79 (18.65) | 134.95 (23.90)
  Week 11 Time 2: number analyzed (Participants) | 22 | 14 | 22
  Week 11 Time 2 | 129.73 (16.59) | 125.71 (12.13) | 136.18 (16.28)
  Week 12 Time 1: number analyzed (Participants) | 21 | 13 | 22
  Week 12 Time 1 | 131.57 (15.10) | 125.54 (15.64) | 140.32 (18.56)
  Week 12 Time 2: number analyzed (Participants) | 21 | 13 | 21
  Week 12 Time 2 | 129.67 (18.11) | 131.85 (14.28) | 134.62 (11.38)

4. Secondary Outcome: Blood Pressure- Diastolic
Description: Blood Pressure is taken for safety reasons
Time Frame: 2 times a week for 12 weeks
Population: Data are reported for those that were measured at each assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 26 | 24 | 26
mmHg
  Week 1 Time 1: number analyzed (Participants) | 26 | 24 | 24
  Week 1 Time 1 | 77.42 (11.61) | 78.75 (9.71) | 79.54 (7.55)
  Week 1 Time 2: number analyzed (Participants) | 24 | 20 | 25
  Week 1 Time 2 | 79.13 (8.04) | 75.75 (11.80) | 80.88 (10.53)
  Week 2 Time 1: number analyzed (Participants) | 25 | 21 | 26
  Week 2 Time 1 | 76.68 (10.48) | 76.48 (15.37) | 79.00 (10.99)
  Week 2 Time 2: number analyzed (Participants) | 24 | 20 | 24
  Week 2 Time 2 | 77.46 (9.07) | 80.70 (11.85) | 79.42 (10.70)
  Week 3 Time 1: number analyzed (Participants) | 24 | 19 | 26
  Week 3 Time 1 | 79.00 (9.04) | 78.79 (10.99) | 78.31 (10.39)
  Week 3 Time 2: number analyzed (Participants) | 22 | 16 | 23
  Week 3 Time 2 | 74.59 (9.59) | 79.50 (11.15) | 78.35 (10.02)
  Week 4 Time 1: number analyzed (Participants) | 24 | 17 | 24
  Week 4 Time 1 | 77.75 (10.61) | 81.88 (13.37) | 80.08 (8.67)
  Week 4 Time 2: number analyzed (Participants) | 23 | 15 | 23
  Week 4 Time 2 | 76.09 (10.87) | 81.67 (12.12) | 80.13 (10.07)
  Week 5 Time 1: number analyzed (Participants) | 23 | 17 | 24
  Week 5 Time 1 | 78.87 (11.29) | 81.41 (10.45) | 80.13 (8.27)
  Week 5 Time 2: number analyzed (Participants) | 21 | 17 | 22
  Week 5 Time 2 | 76.48 (9.28) | 76.53 (12.17) | 80.36 (7.19)
  Week 6 Time 1: number analyzed (Participants) | 23 | 16 | 23
  Week 6 Time 1 | 78.96 (9.15) | 80.63 (13.08) | 80.57 (10.12)
  Week 6 Time 2: number analyzed (Participants) | 22 | 14 | 23
  Week 6 Time 2 | 77.77 (9.13) | 80.43 (10.45) | 83.22 (9.33)
  Week 7 Time 1: number analyzed (Participants) | 22 | 16 | 23
  Week 7 Time 1 | 79.05 (9.92) | 132.31 (200.73) | 79.83 (10.06)
  Week 7 Time 2: number analyzed (Participants) | 22 | 15 | 22
  Week 7 Time 2 | 79.05 (10.82) | 80.00 (11.03) | 81.09 (10.92)
  Week 8 Time 1: number analyzed (Participants) | 21 | 16 | 22
  Week 8 Time 1 | 80.43 (9.72) | 79.50 (8.63) | 81.82 (8.58)
  Week 8 Time 2: number analyzed (Participants) | 20 | 14 | 21
  Week 8 Time 2 | 76.90 (10.23) | 82.71 (14.70) | 82.48 (8.61)
  Week 9 Time 1: number analyzed (Participants) | 22 | 15 | 22
  Week 9 Time 1 | 102.64 (129.67) | 74.67 (12.82) | 81.27 (7.75)
  Week 9 Time 2: number analyzed (Participants) | 21 | 14 | 22
  Week 9 Time 2 | 74.86 (9.24) | 83.50 (7.80) | 80.23 (9.89)
  Week 10 Time 1: number analyzed (Participants) | 22 | 16 | 21
  Week 10 Time 1 | 78.32 (9.18) | 78.75 (12.87) | 81.71 (12.49)
  Week 10 Time 2: number analyzed (Participants) | 21 | 14 | 21
  Week 10 Time 2 | 76.19 (7.49) | 77.57 (10.61) | 76.81 (8.02)
  Week 11 Time 1: number analyzed (Participants) | 22 | 14 | 21
  Week 11 Time 1 | 80.95 (9.32) | 80.57 (12.18) | 85.05 (13.60)
  Week 11 Time 2: number analyzed (Participants) | 22 | 14 | 22
  Week 11 Time 2 | 76.36 (13.17) | 75.36 (22.30) | 82.91 (12.50)
  Week 12 Time 1: number analyzed (Participants) | 21 | 13 | 22
  Week 12 Time 1 | 79.76 (10.72) | 81.46 (8.92) | 84.00 (10.87)
  Week 12 Time 2: number analyzed (Participants) | 21 | 13 | 21
  Week 12 Time 2 | 74.90 (12.48) | 80.15 (10.79) | 84.05 (9.60)

5. Secondary Outcome: CANTAB RVIP Measure: RVP A
Description: RVIP is a computerized measure of attention. This is given at baseline and every 4 weeks over the course of the 12-week study. RVP A' (aka RVIP A PRIME): is a signal detection measure of target sensitivity (i.e., successful response to targets and withholding of responses to non-targets). Range of 0 to 1. Higher scores are better.
Time Frame: Baseline and 12 Weeks
Population: complete case analysis at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 17 | 12 | 15
units on a scale
  Baseline | .86 (.06) | .86 (.05) | .85 (.08)
  Week 12 | .88 (.07) | .84 (.12) | .87 (.08)

6. Secondary Outcome: CANTAB RVIP Measure: RVP B
Description: RVIP is a computerized measure of attention. This is given at baseline and every 4 weeks over the course of the 12-week study. RVP B": A measure of response bias (i.e., bias towards under-responding (to targets) versus over-responding (i.e., to non-targets)) range from -1 to +1, respectively.
Time Frame: Baseline and 12 Weeks
Population: complete case analysis at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 17 | 12 | 15
units on a scale
  Baseline | .77 (.42) | .91 (.13) | .77 (.22)
  Week 12 | .77 (.42) | .91 (.13) | .77 (.22)

7. Secondary Outcome: CANTAB RVIP Measure: RVP FALSE ALARM
Description: RVIP is a computerized measure of attention. This is given at baseline and every 4 weeks over the course of the 12-week study. RVP FALSE ALARM is probability of false alarm. False alarms are responses to non-targets. Higher numbers are worse (i.e., could be seen as a measure of poor response inhibition). Scores range from 0-1 where 1 is the least desirable probablity.
Time Frame: Baseline and 12 Weeks
Population: complete case analysis at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 17 | 12 | 15
units on a scale
  Baseline | .04 (.08) | .01 (.02) | .03 (.04)
  Week 12 | .03 (.03) | .03 (.04) | .02 (.02)

8. Secondary Outcome: CANTAB SST- SSRT
Description: This is the CANTAB SST measure which evaluates response inhibition. Stop Signal Reaction Time (SSRT): The estimate of the length of time between the go stimulus and the stop stimulus at which the subject is able to successfully inhibit their response on 50% of the trials. Range of scores from 0 to 1500 (unit=milliseconds) and lower scores are 'better'.
Time Frame: Baseline and 12 Weeks
Population: Complete cases analyzed at baseline and 12 weeks.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 17 | 12 | 15
milliseconds
  Baseline | 215.3 (89.9) | 277.2 (142.6) | 244.1 (234.8)
  12 Weeks | 241.9 (140.2) | 267.9 (196.6) | 234.8 (129.2)

9. Secondary Outcome: CANTAB SST- Median Correct
Description: This is the CANTAB SST measure which evaluates response inhibition. Stop Signal Reaction Time (SSRT): The estimate of the length of time between the go stimulus and the stop stimulus at which the subject is able to successfully inhibit their response on 50% of the trials. Range of scores from 0 to 1500 (unit=milliseconds) and lower scores are 'better'. Median correct is the median of response times across 'go' trials where the subject has responded on the correct button (right or left).
Time Frame: Baseline and 12 Weeks
Population: Complete cases analyzed at baseline and 12 weeks.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 17 | 12 | 15
milliseconds
  Baseline | 706.3 (260.0) | 619.7 (285.7) | 680.0 (631.5)
  12 Weeks | 608.6 (201.6) | 669.7 (323.5) | 631.5 (150.6)

10. Secondary Outcome: CANTAB SST- SD Correct
Description: This is the CANTAB SST measure which evaluates response inhibition. Stop Signal Reaction Time (SSRT): The estimate of the length of time between the go stimulus and the stop stimulus at which the subject is able to successfully inhibit their response on 50% of the trials. Range of scores from 0 to 1500 (unit=milliseconds) and lower scores are 'better'. SD Correct is the standard deviation of response times across 'go' trials where the subject has responded on the correct button (right or left).
Time Frame: Baseline and 12 Weeks
Population: Complete cases analyzed at baseline and 12 weeks.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 17 | 12 | 15
milliseconds
  Baseline | 276.5 (138.5) | 302.3 (174.6) | 363.4 (214.4)
  12 Weeks | 337.8 (262.9) | 410.6 (276.1) | 492.6 (530.5)

11. Secondary Outcome: Stroop- RT Correct Neutral
Description: Drug Stroop Task is a computerized task which presents words either cocaine-related ('drug') words or non-drug-related ('neutral') words written in colored font. The subject is asked to press a button to indicate the color of the font as quickly and accurately as possible. The task is thought to measure attentional bias to drug-related stimuli. RT Correct Neutral is the mean response time to neutral trials where the subject pressed the correct color response.
Time Frame: weeks 0, 4, 8, 12, 16, 24, 36
Population: Data are reported for those that were assessed at each visit.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 29 | 28 | 28
milliseconds
  Baseline | 785.18 (183.55) | 805.24 (158.88) | 871.07 (191.15)
  Week 4: number analyzed (Participants) | 19 | 15 | 21
  Week 4 | 821.37 (202.21) | 813.66 (182.02) | 845.66 (164.98)
  Week 8: number analyzed (Participants) | 18 | 14 | 19
  Week 8 | 817.69 (220.50) | 741.33 (169.06) | 830.22 (175.45)
  Week 12: number analyzed (Participants) | 17 | 14 | 16
  Week 12 | 764.53 (182.65) | 756.00 (134.75) | 816.47 (180.70)
  Week 16: number analyzed (Participants) | 12 | 9 | 9
  Week 16 | 849.17 (274.21) | 802.90 (219.22) | 895.03 (136.86)
  Week 24: number analyzed (Participants) | 12 | 7 | 9
  Week 24 | 814.09 (255.82) | 769.47 (191.59) | 876.61 (230.52)
  Week 36: number analyzed (Participants) | 8 | 4 | 7
  Week 36 | 824.54 (274.04) | 747.65 (99.74) | 989.42 (156.74)

12. Secondary Outcome: Stroop- RT Correct Drug
Description: Drug Stroop Task is a computerized task which presents words either cocaine-related ('drug') words or non-drug-related ('neutral') words written in colored font. The subject is asked to press a button to indicate the color of the font as quickly and accurately as possible. The task is thought to measure attentional bias to drug-related stimuli. RT Correct Drug is the mean response time to drug trials where the subject pressed the correct color response.
Time Frame: weeks 0, 4, 8, 12, 16, 24, 36
Population: Data are reported for those that were assessed at each visit.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 29 | 28 | 28
milliseconds
  Baseline | 795.40 (185.18) | 806.57 (159.26) | 872.44 (190.94)
  Week 4: number analyzed (Participants) | 19 | 15 | 21
  Week 4 | 825.09 (203.50) | 815.97 (182.08) | 846.59 (165.73)
  Week 8: number analyzed (Participants) | 18 | 14 | 19
  Week 8 | 819.39 (221.27) | 741.46 (168.87) | 829.90 (175.51)
  Week 12: number analyzed (Participants) | 17 | 14 | 16
  Week 12 | 766.90 (181.53) | 755.87 (135.32) | 817.91 (180.55)
  Week 16: number analyzed (Participants) | 12 | 9 | 9
  Week 16 | 847.89 (272.23) | 802.33 (217.92) | 894.15 (136.44)
  Week 24: number analyzed (Participants) | 12 | 7 | 9
  Week 24 | 812.65 (254.72) | 768.93 (189.97) | 874.56 (229.66)
  Week 36: number analyzed (Participants) | 8 | 4 | 7
  Week 36 | 829.28 (278.61) | 747.40 (98.62) | 990.59 (156.20)

13. Secondary Outcome: Stroop- Effect Drug Neutral Mean Correct
Description: Drug Stroop Task is a computerized task which presents words either cocaine-related ('drug') words or non-drug-related ('neutral') words written in colored font. The subject is asked to press a button to indicate the color of the font as quickly and accurately as possible. The task is thought to measure attentional bias to drug-related stimuli. Stroop Effect is difference in response time to drug versus neutral trials (i.e., RT Correct Drug - RT Correct Neutral). A larger stroop effect is 'worse' (thought to indicate more attentional bias to drug related stimuli).
Time Frame: weeks 0, 4, 8, 12, 16, 24, 36
Population: Data are reported for those that were assessed at each visit.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 29 | 28 | 28
milliseconds
  Baseline | .22 (10.60) | 1.33 (5.21) | 1.37 (4.09)
  Week 4: number analyzed (Participants) | 19 | 15 | 21
  Week 4 | 3.71 (8.26) | 2.31 (5.83) | 0.92 (3.08)
  Week 8: number analyzed (Participants) | 18 | 14 | 19
  Week 8 | 1.69 (4.24) | 0.13 (3.40) | -0.12 (3.05)
  Week 12: number analyzed (Participants) | 17 | 14 | 16
  Week 12 | 2.36 (6.23) | -0.12 (3.05) | 1.43 (3.81)
  Week 16: number analyzed (Participants) | 12 | 9 | 9
  Week 16 | -1.27 (4.02) | -0.56 (2.77) | -0.87 (4.50)
  Week 24: number analyzed (Participants) | 12 | 7 | 9
  Week 24 | -1.44 (3.31) | -0.53 (2.24) | -2.05 (3.04)
  Week 36: number analyzed (Participants) | 8 | 4 | 7
  Week 36 | 4.73 (5.53) | -0.25 (1.56) | 1.17 (4.11)

14. Secondary Outcome: Digit Span- LDSF
Description: Digit Span Task description: Orally administered (not computerized) task where subjects are read-aloud lists of digits and asked to repeat them in the same order they heard them (Forward condition). Subjects are given a pair of lists for each digit length - and given a point for each list they get entirely correct. If they get at least one out of the two correct for that length, then the researcher gives them another one of a longer length (one digit longer). If they get both wrong at a given length- that task is ended. The task is then repeated with different digit lists to recall, but they are asked to repeat them or in the reverse order that they heard them (Backward condition). Longest Digit Span Forward (LDSF) is the longest digit span a participant gets correct, in the forward condition. Higher scores are better (Scale of 0 to 9).
Time Frame: Baseline and 12 Weeks
Population: Complete cases at 12 weeks were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 22 | 13 | 17
units on a scale
  Baseline | 5.9 (1.7) | 5.7 (1.3) | 6.4 (2.3)
  12 Weeks | 6.5 (1.4) | 6.8 (1.0) | 7.4 (1.2)

15. Secondary Outcome: Digit Span- DSF
Description: Digit Span Task description: Orally administered (not computerized) task where subjects are read-aloud lists of digits and asked to repeat them in the same order they heard them (Forward condition). Subjects are given a pair of lists for each digit length - and given a point for each list they get entirely correct. If they get at least one out of the two correct for that length, then the researcher gives them another one of a longer length (one digit longer). If they get both wrong at a given length- that task is ended. The task is then repeated with different digit lists to recall, but they are asked to repeat them or in the reverse order that they heard them (Backward condition). Digit Span Forward (DSF) is the number of digit span trials participants got correct in the forward condition. Higher scores are better (Scale of 0 to 14).
Time Frame: Baseline and 12 Weeks
Population: Complete cases at 12 weeks were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 22 | 13 | 19
units on a scale
  Baseline | 9.3 (3.0) | 9.9 (2.3) | 10.7 (2.1)
  12 Weeks | 10.5 (2.6) | 10.7 (1.8) | 11.2 (3.1)

16. Secondary Outcome: Digit Span- LDSB
Description: Digit Span Task description: Orally administered (not computerized) task where subjects are read-aloud lists of digits and asked to repeat them in the same order they heard them (Forward condition). Subjects are given a pair of lists for each digit length - and given a point for each list they get entirely correct. If they get at least one out of the two correct for that length, then the researcher gives them another one of a longer length (one digit longer). If they get both wrong at a given length- that task is ended. The task is then repeated with different digit lists to recall, but they are asked to repeat them or in the reverse order that they heard them (Backward condition). Longest Digit Span Backward (LDSB) is the longest digit span participants got correct, in the backward condition. Higher scores are better (Scale of 0 to 8).
Time Frame: Baseline and 12 Weeks
Population: Complete cases at 12 weeks were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 22 | 13 | 17
units on a scale
  Baseline | 4.2 (1.7) | 3.2 (0.9) | 4.0 (1.7)
  12 Weeks | 4.2 (1.2) | 4.3 (1.4) | 3.9 (1.6)

17. Secondary Outcome: Digit Span- DSB
Description: Digit Span Task description: Orally administered (not computerized) task where subjects are read-aloud lists of digits and asked to repeat them in the same order they heard them (Forward condition). Subjects are given a pair of lists for each digit length - and given a point for each list they get entirely correct. If they get at least one out of the two correct for that length, then the researcher gives them another one of a longer length (one digit longer). If they get both wrong at a given length- that task is ended. The task is then repeated with different digit lists to recall, but they are asked to repeat them or in the reverse order that they heard them (Backward condition). Digit Span Forward (DSB) is the number of digit span trials participants got correct in the backward condition. Higher scores are better (Scale of 0 to 14).
Time Frame: Baseline and 12 Weeks
Population: Complete cases at 12 weeks were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine 8mg | Galantamine 16mg | Placebo
Number analyzed (Participants) | 22 | 13 | 19
units on a scale
  Baseline | 8.3 (3.1) | 7.2 (1.5) | 7.6 (1.9)
  12 Weeks | 8.3 (2.1) | 8.5 (2.7) | 7.3 (2.7)

ADVERSE EVENTS:
Arm/Group | Placebo | Galantamine 8mg | Galantamine 16mg
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 19/32 | 13/31 | 15/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | Galantamine 8mg (N=31) | Galantamine 16mg (N=30)
Confusion (Psychiatric disorders) | 1 | 1 | 2
Hallucinations (Psychiatric disorders) | 0 | 1 | 1
Delusions (Psychiatric disorders) | 0 | 0 | 2
Agitation (Psychiatric disorders) | 5 | 3 | 4
Tiredness (General disorders) | 7 | 6 | 8
Drowsiness (General disorders) | 0 | 1 | 2
Insomnia (General disorders) | 5 | 1 | 5
Nightmares (General disorders) | 2 | 0 | 2
Irresponsible Behavior (Psychiatric disorders) | 2 | 0 | 1
Depression (Psychiatric disorders) | 0 | 3 | 3
Anxiety (Psychiatric disorders) | 4 | 3 | 4
Tingling (Nervous system disorders) | 1 | 0 | 0
Cramps (Gastrointestinal disorders) | 2 | 1 | 0
Headache (General disorders) | 7 | 2 | 2
Blurred Vision (Eye disorders) | 1 | 2 | 3
Dry Mouth (General disorders) | 2 | 2 | 2
Increased Perspiration (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Flushing (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 5
Urinary Frequency (Renal and urinary disorders) | 3 | 5 | 2
Dizziness (General disorders) | 2 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0 | 3
Increased Appetite (Metabolism and nutrition disorders) | 2 | 1 | 0
Heartburn (Gastrointestinal disorders) | 4 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 1 | 0
Euphoria (Psychiatric disorders) | 0 | 0 | 1
Poor Concentration (General disorders) | 1 | 0 | 0
Chills (Nervous system disorders) | 1 | 1 | 1
Increased Libido (Psychiatric disorders) | 1 | 0 | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0 | 2
Nausea/Vomiting (Gastrointestinal disorders) | 2 | 0 | 2
Disturbed Concetration (General disorders) | 0 | 3 | 3
Decreased Libido (Psychiatric disorders) | 0 | 0 | 1
Fainting (Nervous system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes